CLINICAL TRIAL: NCT07395869
Title: Pain and Itch Neuromodulation: Effects of Offset Analgesia, Placebo, and Nocebo and Topographical Distribution of Itch and Pain Receptors
Brief Title: Off-set Analgesia Induced by Cold Temperature
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Associate Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20250017 Project 1
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- off-set analgesia (Experimental): The tests of off-set analgesia will be performed using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device. Two protocols will be applied: heat off-set analgesia and cold off-set analgesia.
  Interventions: Other: Heat off-set analgesia; Other: Cold off-set analgesia

INTERVENTIONS:
Other: Heat off-set analgesia — The tests of off-set analgesia will be performed using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Other: Cold off-set analgesia — The tests of off-set analgesia will be performed using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device.

SUMMARY:
In this study, it will be investigated if the phenomenon of offset analgesia, usually associated with painful heat stimulation, could also be induced using cold painful temperatures.

DETAILED DESCRIPTION:
After filling some questionnaires, two areas (4x4 cm, 4 cm apart) will be selected on each forearm of the subjects. The areas will be randomly treated with one of the following trials: hot experimental trial, hot control trial, cold experimental trial, and cold control trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other drugs
* Previous or current history of neurological, immunological, musculoskeletal, cardiac disorder or psychiatric diagnoses that may affect the results (e.g., neuropathy, muscular pain in the upper extremities, anxiety, depression, schizophrenia, etc.)
* Moles, wounds, scars, or tattoos in the area to be treated or tested
* Current use of medications that may affect the trial such as antihistamines and pain killers
* Skin diseases
* Consumption of alcohol or painkillers 24 hours before the study days and between these
* Acute or chronic pain and itch
* Participation in other trials within 1 week of study entry (4 weeks in the case of pharmaceutical studies)
* Contraindications to capsaicin, including intolerance to chili or burns or wounds at the application site (sub-project 4 only)
* The subject is assessed as unable to engage in the necessary cooperation required by the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Measuring pain by computerized Visual Analog Scale Scoring | Immediately after the intervention
  We will ask the subjects to rate the sensation of pain on a 100

SECONDARY OUTCOMES:
Pain Catastrophizing Scale (PCS). | Baseline
  The PCS assesses negative and exaggerated coping concerning anticipated or experienced painful stimuli. Thirteen items have to be answered on a 5-point Likert-type scale ranging from 0 (Not at all) to 4 (all the time).
Learned Helplessness Scale (LHS) | Baseline
  The questionnaire consists of 20 items, and the participant's response to each item is rated on a 4-point Likert scale branging from strongly agree (1) to strongly disagree (4).
Depression, Anxiety, Stress Scale (DASS-21) | Baseline
  The questionnaire measures the magnitude of depression, anxiety, and stress. Each of these three subscales consists of 7 questions answered using a 0-3 Likert scale, with 0 meaning "it did not apply to me", and 3 meaning "it applied to me very much"
Reinforcement Sensitivity Theory - Personality Questionnaire (RST-PQ). | Baseline
  The RST-PQ contains in total 65 items must be answered on a Response scale: 4-point Likert (Strongly disagree → Strongly agree).
Positive And Negative Affect Schedule (PANAS) | Baseline
  Twenty words are associated with the subject's current feelings and have to be rated on a 5-points Likert-type scale from: Very slightly or not at all to extremely.
Difficulties in Emotion Regulation Scale Short Form (DERS-SF) | Baseline
  The questionnaire is an 18-item measure used to identify emotional regulation issues in adults. Participants rate each item on a 5-point Likert scale (from 1 to 5).
Emotion Regulation Questionnaire (ERQ) | Baseline
  This questionnaire is designed to assess individual differences in the habitual use of two emotion regulation strategies: cognitive reappraisal and expressive suppression. Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree), where 4 means (neutral).

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Neuroplasticity and Pain Faculty of Medicine, Aalborg University Selma Lagerløfs Vej 249 9260 Gistrup, Denmark, Aalborg, Aalborg, Denmark